CLINICAL TRIAL: NCT00614458
Title: 10493 - MK-0518 Intensification and HDAC Inhibition in Depletion of Resting CD4+ T Cell HIV Infection
Brief Title: MK-0518 Intensification And HDAC Inhibition In Depletion Of Resting CD4+ T Cell HIV Infection
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to insufficient funds
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Abbott (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, David Margolis, MD, Principal Investigator, University of North Carolina, Chapel Hill
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10493; R01AI064074 (NIH); P30AI050410 (NIH); U01AI067854 (NIH); NCT00576290 (obsolete NCT alias)
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Results first posted 2011-10-25 (Estimated); Last update posted 2011-10-25 (Estimated); Status verified 2011-09

CONDITIONS: HIV Infections
Keywords: latent HIV; resting CD4+ T cell; valproic acid (VPA); Raltegravir (MK-0518) intensification; HIV replication; treatment experienced
MeSH Terms: conditions — HIV Infections | interventions — Raltegravir Potassium; Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Raltegravir and VPA to ART (Experimental): raltegravir 400mg po BID; valproic acid 1000mg - 2000mg daily
  Interventions: Drug: Raltegravir; valproic acid

INTERVENTIONS:
Drug: Raltegravir; valproic acid — raltegravir 400mg po BID; valproic acid 1000mg - 2000mg daily
  Other Names: raltegravir (MK 0518); Valproic acid (VPA) (depakote)

SUMMARY:
The purpose of this research study is to see if HIV that persists despite current antiviral therapy can be targeted by new treatments. We will see if adding Raltegravir (MK-0518) and Valproic acid (VPA) to current ART can decrease the amount of latent HIV.

DETAILED DESCRIPTION:
The purpose of this research study is to see if HIV that persists despite current antiviral therapy can be targeted by new treatments. Eradicating this hidden, persistent virus (which we will call "latent HIV") may some day allow HIV to be eliminated from an infected person. Recently it has been discovered that a class of medicines, called histone deacetylase (HDAC) inhibitors, may cause the HIV that hides within some of the cells of your body to be expressed ("unmasked"). The HDAC inhibitor we will use in this study to unmask or flush out the latent HIV within your cells is called valproic acid (VPA) and is commonly used to treat seizures and depression under the brand name Depakote. VPA has been safely given to people with HIV for the treatment of seizures or depression.

In our first study, we recruited 4 volunteers with HIV-1 infection taking antiviral therapy in whom there were <50 copies/ml (undetectable) of HIV virus RNA in their blood for over 6 months. In addition to continuing their anti-HIV medications, we started them on Fuzeon, a new injected anti-HIV medication, for one month. We then added VPA to the anti-HIV medications and Fuzeon for 3 months. At the end of the study, we found that latent HIV was significantly decreased. No safety problems with VPA and antiviral medicines were noted. However, having initiated Fuzeon and VPA simultaneously we could not determine with confidence that our findings were due to the effect of VPA alone.

In the next study we added VPA to the therapy of patients taking standard antiretroviral therapy (ART). Eight patients have been studied so far, but only three have yet had a significant decrease in latent HIV. It may be that VPA does not work in everyone, or that stronger HIV therapy is needed in some people to drain latent HIV. And in a different study, no decrease at all was found in the number of infected cells in people taking ART who were prescribed valproate for other reasons.

In this study, we wish to add a different new anti-HIV medicine, which is a pill, Raltegravir (MK-0518). Raltegravir blocks the virus from permanently entering the DNA of your T cells, and so is called an integrase inhibitor. Raltegravir is investigational. This means the U.S. Food and Drug Administration (FDA) have not yet approved it for sale. We will see if adding Raltegravir and VPA to your current ART can decrease the amount of latent HIV. If adding Raltegravir and VPA to your ART has no effect, you will have reached the end of the study. If adding Raltegravir and VPA decreases latent infection, we will stop VPA but continue Raltegravir to see if this new integrase inhibitor decreases latent infection. This study does not expect to cure your HIV, but only to take the first step towards that far-away goal.

You are asked to join this study because you are infected with the HIV-1 virus; you are 18 years of age; you are able and willing to sign an informed consent.; you are able to have laboratory tests within the study specific criteria; and you have adequate vein access for leukopheresis.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection
* Men and women age ≥18 years.
* Ability and willingness of subject or legal guardian/representative to give written informed consent.
* Karnofsky performance status >70.
* Willing to adhere to protocol therapy and judged adherent to antiretroviral therapy, and can comply with time requirements for protocol-specified visits and evaluations.
* On potent antiretroviral therapy, defined as at least 2 nucleoside reverse transcriptase inhibitors (NRTIs) plus at least 1 protease inhibitor (PI) or non-nucleoside reverse transcriptase inhibitor (NNRTI), without changes in the 24 weeks immediately prior to entry. Prior changes in or elimination of medications for easier dosing schedule, intolerance, or toxicity are permitted.
* Have no contraindications to valproic acid (VPA) therapy (pregnancy, bleeding disorders, history of pancreatitis, history of hepatitis).
* Have adequate vascular access for leukopheresis
* Plasma HIV-1 RNA never > 50 copies/ml on two consecutive occasions for ≥ 6 months.
* CD4 cell count > 300 cells/µl.
* Screening serum fasting glucose below 120 mg/dl, creatinine no more than 1.5 times the upper limit of the normal range, serum AST, ALT, and total bilirubin less than 2 times the upper limit of the normal range, and fasting triglycerides < 400mg/dl.
* Female study volunteers who are not of reproductive potential or whose male partner(s) has undergone successful vasectomy with documented azoospermia or has documented azoospermia for any other reason, are eligible without requiring the use of contraception.
* All women of reproductive potential must have a negative urine beta-HCG pregnancy test performed at screening, day 0, week 4, week 8, week 12, and every scheduled study visit thereafter.
* All study volunteers must agree not to participate in a conception process and, if participating in sexual activity that could lead to pregnancy, the female study volunteer/male partner must use two reliable methods of contraception simultaneously while receiving the protocol-specified medications and for 6 weeks after stopping the medications. Subjects must use a reliable barrier method of contraception along with another form of contraception. For women receiving ritonavir, estrogen-based contraceptives are not reliable and an alternative method should be used.

Exclusion Criteria:

* Receiving zidovudine (AZT). Due to the inhibition of zidovudine metabolism mediated by Valproic acid (VPA) a theoretical increase risk of zidovudine-induced anemia exists.
* Using drugs known to interact with valproate or raltegravir (MK-0518)
* Pregnant or nursing.
* Anemic (Hemoglobin < 10gm/dl)
* Seropositive for hepatitis C RNA or hepatitis B surface antigen within 90 days prior to entry.
* Have signs or symptoms of hepatic decompensation
* Received blood transfusions or hematopoetic growth factors within 90 days.
* Use of any of the following within 90 days prior to entry: systemic cytotoxic chemotherapy, investigational agents, immunomodulators.
* Active drug or alcohol use or dependence.
* Serious illness requiring systemic treatment or hospitalization until subject either completes therapy or has been clinically stable on therapy, in the opinion of the site investigator, for at least 90 days prior to entry.
* Compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric illness or a physical illness, e.g., infectious disease.
* Treatment for an active AIDS-defining opportunistic infection within 90 days prior to screening.

For this pilot study of no direct benefit to subjects, non-English speaking patients are excluded. In the future, if this study is expanded to include a larger sample size, this exclusion criterion may be removed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2007-04; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David M Margolis, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Result] Archin NM, Cheema M, Parker D, Wiegand A, Bosch RJ, Coffin JM, Eron J, Cohen M, Margolis DM. Antiretroviral intensification and valproic acid lack sustained effect on residual HIV-1 viremia or resting CD4+ cell infection. PLoS One. 2010 Feb 23;5(2):e9390. doi: 10.1371/journal.pone.0009390. PMID 20186346

RESULTS

PARTICIPANT FLOW:
Groups:
- Effect on Latent HIV of Adding Raltegravir and VPA to ART: Single arm pilot study that measured the effect of adding Raltegravir and Valproic acid (VPA) and current antiretroviral therapy (ART) on the persistence of latent HIV infection within circulating, resting CD4+ T cells in patients stably suppressed by ART
Period: Overall Study
Arm/Group | Effect on Latent HIV of Adding Raltegravir and VPA to ART
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Effect on Latent HIV of Adding Raltegravir and/or VPA to ART: Single arm pilot study that measured the effect of adding Raltegravir and/or VPA and current ART on the persistence of latent HIV infection within circulating, resting CD4+ T cells in patients stably suppressed by ART
Arm/Group | Effect on Latent HIV of Adding Raltegravir and/or VPA to ART
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 36 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: A Change in the Number of HIV Infected Cells.
Description: A change in infected cells from prior to the initiation of VPA and MK0518 to after 20 weeks of treatment.
Time Frame: 20 weeks
Population: All participants analyzed per protocol
Measure: Median (95% Confidence Interval); unit: infected cells /million cells
Arm/Group | Effect on Latent HIV of Adding Raltegravir and VPA to ART
Number analyzed (Participants) | 6
infected cells /million cells | 0.390 [0.03 to 10]

ADVERSE EVENTS:
Arm/Group | Effect on Latent HIV of Adding Raltegravir and/or VPA to ART
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No